CLINICAL TRIAL: NCT05201339
Title: Effect of Head-neck Rotation on the Success Rate At First Attempt of I-gel™ Insertion
Brief Title: Effect of Head-neck Rotation on I-gel™ Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Karam Nam, MD, Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LMA_HNRotation
Record Dates: First submitted 2021-12-21; First posted 2022-01-21 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Supraglottic Airway Device; Intubation; Difficult or Failed; Airway Complication of Anesthesia
Keywords: Supraglottic airway device; Intubation; Airway

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard method (Active Comparator): Insert I-gel™ according to the manufacturer's instruction. Take the sniffing position and gently move the i-gel™ along the hard palate to the soft palate and the posterior oropharynx.
  Interventions: Procedure: Standard method
- Head-neck rotation (Experimental): After rotating the patient's head and neck to the left maximally, insert the i-gel™ from the right side of the tongue to the midline. When the tip reaches the soft palate and oropharynx positions, turn the head and neck back to the neutral position.
  Interventions: Procedure: Hean and Neck Rotation

INTERVENTIONS:
Procedure: Standard method — Insert I-gel™ according to the manufacturer's instruction. Take the sniffing position and gently move the i-gel™ along the hard palate to the soft palate and the posterior oropharynx.
  Arms: Standard method
Procedure: Hean and Neck Rotation — After rotating the patient's head and neck to the left maximally, insert the i-gel™ from the right side of the tongue to the midline. When the tip reaches the soft palate and oropharynx positions, turn the head and neck back to the neutral position.
  Arms: Head-neck rotation

SUMMARY:
According to previous studies, head and neck rotation reduces the tongue from being rolled back by gravity, which resulted in increasing patency of the upper airway. Therefore, the purpose of this study is to verify whether head and neck rotation increases the first attempt success rate of i-gel™.

DETAILED DESCRIPTION:
I-gel™ insertion has been reported that the success rate of insertion on the first attempt is 78.5%. There may be several causes of insertion failure. Tongue folding is a major obstacle preventing appropriate i-gel™ placement. To solve this problem, the previous study has proven the efficacy of the rotational technical for I-gel™ insertion and reported a success rate of 97%.

However, the rotation of i-gel™ in the oral cavity may be limited, and it may take some learning curve to get used to it. According to previous studies, head and neck rotation increases the cross-sectional area of the upper airway, which resulted in increasing patency of the upper airway. Therefore, the purpose of this study is to verify whether head and neck rotation increases the first attempt success rate of i-gel™.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status Classification Grade 1-3
* Patients who can provide written consent to participate in clinical trials
* Patients requiring the I-gel™ during surgery

Exclusion Criteria:

* Outpatient surgery
* Patients who have the neurologic disease or cognitive impairment
* Patients who take antipsychotic drugs
* Body mass index > 35 kg/m2
* Mouth opening < 2.5 cm
* Limited neck extension or cervical mobilization (Ex: Atlanto-axial subluxation, History of cervical spine surgery or head and neck surgery)
* Those with a recent sore throat
* Those with weak dentation
* Patients at risk of aspiration (Ex: Pregnancy, Gastroesophageal reflux disease or hiatus hernia)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | Induction of anesthesia during intraoperative period
  After the first attempt on insertion of i-gel™ without withdrawal or redirection, the effectiveness of the airway is judged based on a square-wave capnograph and no audible leak with peak airway pressures ≥ 10 cmH2O during manual ventilation.

SECONDARY OUTCOMES:
Second attempt success rate | Induction of anesthesia during intraoperative period
  After the second attempt on insertion of i-gel™, the effectiveness of the airway is judged based on a square-wave capnograph and no audible leak with peak airway pressures ≥ 10 cmH2O during manual ventilation.
Insertion time for successful insertion; s | Induction of anesthesia during intraoperative period
  Time from insertion of i-gel™ into the oral cavity until appropriate placement.
Time required for successful insertion; s | Induction of anesthesia during intraoperative period
  Time insertion of i-gel™ into the oral cavity until After the first attempt on insertion of i-gel™ without withdrawal or redirection, the effectiveness of the airway is judged based on a square-wave capnograph and no audible leak with peak airway pressures ≥ 10 cmH2O during manual ventilation.
Third attempt | Induction of anesthesia during intraoperative period
  If the attempt of assigned method fails twice, then try third attempt.
Third attempt success rate | Induction of anesthesia during intraoperative period
  If the attempt of assigned method fails, but the third attempt is successful with another method.
Manipulations required rate | Induction of anesthesia during intraoperative period
  An assistant assists when all attempt fail.
Change to intubation | Induction of anesthesia during intraoperative period
  Conversion rate from insertion of i-gel™ to tracheal intubation.
Blood staining after extubation | Induction of anesthesia during intraoperative period
  Blood stating to evaluate the postoperative complication and outcome in patients received each intubation method during surgery
Sore throat after extubation | Extubation during intraoperative period
  Sore throat to evaluate the postoperative complication and outcome in patients received each intubation method during surgery
Hoarseness after extubation | Extubation during intraoperative period
  Hoarseness to evaluate the postoperative complication and outcome in patients received each intubation method during surgery
Sore throat at 24 hours after surgery | 24 hours after surgery (up to 24hours)
  Sore throat to evaluate the postoperative complication and outcome in patients received each intubation method during surgery
Hoarseness at 24 hours after surgery | 24 hours after surgery (up to 24hours)
  Hoarseness to evaluate the postoperative complication and outcome in patients received each intubation method during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karam Nam, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Nam K, Park SJ, Ju JW, Cho YJ, Jeon Y. Comparison between head rotation and standard techniques for i-gel insertion: a randomized controlled trial. BMC Anesthesiol. 2024 Jul 10;24(1):229. doi: 10.1186/s12871-024-02621-7. PMID 38987667